CLINICAL TRIAL: NCT00325806
Title: Prevention of Hypertension in Patients With High-Normal Blood Pressure With the Angiotensin-Converting-Enzyme-Inhibitor Ramipril - a Randomised Prevention Trial of the German Hypertension League.
Brief Title: Ramipril - Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE498_3E03
Record Dates: First submitted 2006-04-11; First posted 2006-05-15 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
Primary objective:

Mean values of systolic and diastolic office blood pressure

Secondary objectives:

Total mortality, occurrence of cardio- and cerebrovascular events, change of mean blood pressure (ABPM : Ambulatory Blood Pressure Monitoring) during the observation

ELIGIBILITY:
Inclusion Criteria:

* no previous antihypertensive therapy
* high-normal blood pressure according to the JNC-VI definition (systolic 130 - 139 and/or diastolic 85 - 89 mmHg)

Exclusion Criteria:

* antihypertensive therapy
* blood pressure greater 140/90 mmHg or ABPM greater 135/85 mmHg

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2000-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Mean systolic and diastolic 24-hour blood pressure in ABPM

SECONDARY OUTCOMES:
Overall mortality and total number of cardiovascular and cerebro-vascular events
Changes in mean blood pressure readings over time
Reasons for admissions to hospital/-stays
Occurrence of pathological fasting glucose levels in serum/pathological HbA1c levels.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

REFERENCES:
- [Result] Luders S, Schrader J, Berger J, Unger T, Zidek W, Bohm M, Middeke M, Motz W, Lubcke C, Gansz A, Brokamp L, Schmieder RE, Trenkwalder P, Haller H, Dominiak P; PHARAO Study Group. The PHARAO study: prevention of hypertension with the angiotensin-converting enzyme inhibitor ramipril in patients with high-normal blood pressure: a prospective, randomized, controlled prevention trial of the German Hypertension League. J Hypertens. 2008 Jul;26(7):1487-96. doi: 10.1097/HJH.0b013e3282ff8864. PMID 18551027